CLINICAL TRIAL: NCT02504398
Title: A Randomized Controlled Trial of Injection Technique for Infant Vaccination
Brief Title: Speed of Injection and Pain During Routine Infant Vaccinations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31803
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Routine Infant Immunizations; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast injection (Experimental): Vaccine injections will be given at a rate of approximately 2-4 ml/sec by the immunizer
  Interventions: Other: Fast injection speed by immunizer
- Slow injection (Active Comparator): Vaccine injections will be given at a rate of approximately 10 ml/sec by the immunizer
  Interventions: Other: Slow injection speed by immunizer

INTERVENTIONS:
Other: Fast injection speed by immunizer
  Arms: Fast injection
Other: Slow injection speed by immunizer
  Arms: Slow injection

SUMMARY:
Vaccine injections are a significant source of pain for infants. Altering the injection speed when administering vaccines may be an effective intervention and is feasible (cost neutral). At present, there are no data regarding impact of injection speed on vaccine injection pain in infants. The aim of this study is to address this knowledge gap and to compare the impact of slow and fast vaccine injection speeds on pain during routine infant vaccinations.

DETAILED DESCRIPTION:
To date, there has been no evidence-based guidance regarding the rate at which vaccines should be injected to minimize pain. This has led to a disparity in practice. Some vaccinators favour a slow rate of injection (around 8-10 sec/mL) while others prefer a more rapid rate of injection (around 2-4 sec/mL).The slow injection method leads to a longer needle dwelling time with the increased possibility of the needle moving around and causing pain by damaging muscle tissue. Rapid injection, on the other hand, may lead to a sudden distension of muscle tissue, which itself could be painful. Allowing the muscle sufficient time to distend in order to accommodate the vaccine might minimize pain. This study will address the identified knowledge gap by comparing pain in infants undergoing routine vaccinations with a fast vs. slow injection speed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2 and 4 month old infants receiving their primary vaccine injections, PediacelTM (0.5mL) and PrevnarTM (0.5mL) (in conjunction with and preceded by oral RotarixTM vaccine) and healthy 6 month old infants receiving their routine vaccine injection, PediacelTM (0.5mL)

Exclusion Criteria:

* Infants with impaired neurological development; history of seizures; administration of sedatives or narcotics in the preceding 24 hours; parental inability to use study tools; parent vaccine refusal; prior participation in the trial; and refusal to be video recorded

Ages: 2 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Infant Behavioural Pain Score | up to 1 minute post-vaccinations
  Assessed using the Modified Behavioural Pain Scale (0-10) from videotapes of the procedure

SECONDARY OUTCOMES:
Infant Parent-rated Pain Score | up to 2 minutes
  Assessed using a Numerical Rating Scale (0-10) by parent in real time
Infant Cry duration | up to 2 minutes
  Assessed in 1 minute intervals for 2 minutes following vaccinations from videotapes

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Pediatric Consultants, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taddio A, Wong H, Welkovics B, Ilersich AL, Cole M, Goldbach M, Ipp M. A randomized trial of the effect of vaccine injection speed on acute pain in infants. Vaccine. 2016 Sep 7;34(39):4672-4677. doi: 10.1016/j.vaccine.2016.08.023. Epub 2016 Aug 12. PMID 27527817